CLINICAL TRIAL: NCT01928706
Title: Oral Health Related Quality of Life of Edentulous Patients After Relining Mandibular Dentures With Soft and Hard Denture Liners.
Brief Title: Quality of Life After Denture Relining
Acronym: OHRQoL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Marina Xavier Pisani, Dds, MsC, PhD, Fundação de Amparo à Pesquisa do Estado de São Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 24021985
Record Dates: First submitted 2013-08-06; First posted 2013-08-27 (Estimated); Last update posted 2013-08-27 (Estimated); Status verified 2013-08

CONDITIONS: Quality of Life
Keywords: edentulism; denture liner; prosthodontics; OHIP EDENT
MeSH Terms: interventions — kooliner

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Denture liner Mucopren Soft; Group 1 (Experimental): The existing mandibular dentures were relined with a soft silicone-based denture liner (Mucopren Soft; Group 1; n=22).
  Interventions: Other: Denture liner Mucopren Soft; Group 1
- Denture liner Kooliner; Group 2 (Active Comparator): The existing mandibular dentures were relined with a a hard acrylic resin based denture liner (Kooliner; Group 2 n=22).
  Interventions: Other: Denture liner Kooliner; Group 2

INTERVENTIONS:
Other: Denture liner Mucopren Soft; Group 1 — Complete denture wearers had their existing mandibular dentures relined with a soft silicone-based denture liner (Mucopren Soft; Group 1; n=22)
  Other Names: Mucopren Soft relining
  Arms: Denture liner Mucopren Soft; Group 1
Other: Denture liner Kooliner; Group 2 — Complete denture wearers had their existing mandibular dentures relined with a hard acrylic resin based denture liner (Kooliner; Group 2;n=22) with chairside procedures.
  Other Names: Kooliner
  Arms: Denture liner Kooliner; Group 2

SUMMARY:
Purpose: the aim of the present study was to analyze the impact of mandibular denture relining with soft or hard denture liners in the oral health related quality of life (OHRQoL) of edentulous patients.

The null hypothesis was that there would be no difference in OHRQoL findings after mandibular denture relining between patient groups treated with hard or soft denture liners.

DETAILED DESCRIPTION:
Complete denture wearers had their existing mandibular dentures relined with a soft silicone-based denture liner (Mucopren Soft; Group 1; n=22) or a hard acrylic resin based denture liner (Kooliner; Group 2; control n=22) with chairside procedures. The OHIP EDENT (Oral Health Impact profile) questionnaire was given to patients prior to reline procedures (baseline-T0) and 90 days (T90) post relining. Three possible answers and scores were proposed for each question: never (0), sometimes (1) and almost always (2). Results were analyzed by means of the generalized linear model (p≤0.05) considering two factors: time (T0 and T90) and group (hard and soft denture liners).

ELIGIBILITY:
Inclusion Criteria:

* Edentulous in both jaws
* Complete denture wearers
* Clinically acceptable occlusal relationships
* Healthy mucosa, i.e. with no signs of inflammation, traumatic lesions, candidiasis or hyperplasia.

Exclusion Criteria:

* Residual vertical bone height of 10 mm or less
* No attached mucosa in any region of mandible (type E)
* Dentures with deteriorated intaglio surfaces
* Dentures with large pre-existing fractures
* Dentures with severely altered occlusal vertical dimension
* Extremely worn artificial teeth
* Dentures with unsatisfactory occlusions
* Neurological diseases
* Lack of motor coordination
* Difficulty of understanding instructions and the conditions of the study
* Patients with residual roots, cysts or bone spicules
* Patients with allergies to methyl methacrylate or silicone
* Knife-edge mandibular ridges.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-03; Primary Completion 2012-02 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Oral health related quality of life at 90 days after denture relining | The oral health related quality of life was evaluated before relining (T0- baseline), and after 90 days post denture relining.
  The Oral Health Related Quality of Life (OHRQoL) was assessed through the application of the questionnaire OHIP EDENT at baseline and 90 days post denture relining. Four domains developed for the Brazilian OHIP-EDENT9 were used: (D1) 'masticatory-related complaints, (D2) 'psychological discomfort and disability', (D3) 'social disability' and (D4) 'oral pain and discomfort'.
  The questionnaires were carried out via interviews by one individual examiner , who was blinded for the denture liner. The interviews lasted approximately ten minutes.Three possible answers to questions one to nineteen with their scores in parenthesis were given as options: never (0), sometimes (1) or almost always (2).

CONTACTS AND LOCATIONS:
Overall Officials: C H Lovato, pHD, Principal Investigator — Ribeirao Preto Dental School University of Sao Paulo
Locations (1):
- Ribeirao Preto Dental School University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil